CLINICAL TRIAL: NCT00829413
Title: Characterization Of Focal Liver Lesions With Sonovue®-Enhanced Ultrasound Imaging: A Phase III, Intrapatient Comparative Study Versus Unenhanced Ultrasound Imaging Using Histology Or Combined Imaging/Clinical Data As Truth Standard
Brief Title: SonoVue®-Enhanced Ultrasound (US) Versus Unenhanced US for Focal Liver Lesion Characterization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR1-130
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2017-11

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients who received SonoVue (Other): Patients with at least one target lesions requiring work-up for characterization to undergo
  * Unenhanced ultrasound of the target lesion (UE-US): gray scale and Doppler (color or power imaging) ultrasound investigations of the target lesion using commercially available ultrasound equipment and standard techniques (B-mode or Harmonic imaging) to study the anatomy of the target lesion and surrounding parenchyma;
  * SonoVue-enhanced ultrasound of the target lesion (CE-US):procedures described in protocol Section 7.5.1.2, to study the lesion vascularity in comparison to the surrounding parenchyma; and
  * Truth standard
  2.4 mL of sulfur hexafluoride microbubbles (SonoVue®) will be administered as a bolus injection in a peripheral vein.
  Interventions: Drug: SonoVue®

INTERVENTIONS:
Drug: SonoVue® — SonoVue (2.4 mL)
  Other Names: sulfur hexafluoride microbubbles

SUMMARY:
The purpose of this study is to demonstrate the Sensitivity and Specificity of SonoVue®-enhanced ultrasound is superior to that of unenhanced ultrasound for the characterization of benign versus malignant FLLs using final diagnosis based on histology or combined imaging (CE-CT and/or CE MRI)/clinical data as truth standard.

DETAILED DESCRIPTION:
Unit of analysis for the outcome measures was the lesion, equivalent to the subject, since each subject had a single lesion that was to be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Male/female.
* Provides written Informed Consent and is willing to comply with protocol requirements.
* Is at least 18 years of age.
* Has at least 1 FLL (target lesion) requiring work-up for characterization. Target lesions may include those:

Incidentally detected, In subjects with chronic hepatitis or liver cirrhosis, In subjects with known history of malignancy.

* Is scheduled for surgical removal or biopsy of the target lesion from 24 hours to 30 days after the SonoVue® administration OR
* In case tissue biopsy is not indicated nor surgery planned, is scheduled for or has performed a CE-CT and/or CE-MRI of the target lesion from 30 days to 48 hours prior to or from 24 hours to 30 days after the administration of SonoVue®.

Exclusion Criteria:

* Has an acoustic window insufficient for adequate ultrasound examination of the liver.
* Has a FLL that cannot be identified with unenhanced ultrasound.
* Has received or is scheduled for antineoplastic chemotherapy or an invasive procedure in the time period between test procedures and truth standard assessments which may have modified the target lesion.
* Is receiving any other contrast medium, within the 48 hours before and up to 24 hours following the administration of SonoVue®.
* Has previously been enrolled in and completed this study.
* Known right to left cardiac shunt, bidirectional or transient.
* Has any known allergy to 1 or more of the ingredients of the investigational product (sulfur hexafluoride or to any components of SonoVue®).
* Has any contraindication to 1 of the planned imaging procedures (ultrasound, CT or MRI), e.g., implants, claustrophobia, inadequate medical conditions etc.
* Has received an investigational compound within 30 days before admission into this study.
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations.
* Is determined by the Investigator that the subject is clinically unsuitable for the study.
* Is a pregnant or lactating female. Exclude the possibility of pregnancy by:

testing on site at the institution serum βHCG within 24 hours prior to the start of SonoVue® administration, surgical history (e.g., tubal ligation or hysterectomy), post menopausal with a minimum 1 year without menses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Spinazzi, M.D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics Inc., Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date (first subject enrolled): 15 June 2010; Study completion date (last patient completed study related activities): 18 February 2013. The study was conducted at 18 investigational sites; 11 sites throughout the United States (USA), 5 sites in Europe, and 2 sites in Canada.
Pre-assignment Details: A total of 67 patients received SonoVue in the training phase and were included only in safety population. A total of 259 patients received SonoVue in the efficacy phase. The 67 patients, included within the "Not Completed" category below, are the training patients.
Groups:
- Safety Population: Interventions included SonoVue administration, unenhanced (UE-US) and SonoVue-enhanced ultrasound (CE-US) and definitive truth standard diagnosis.
  Any patient who received SonoVue is included in the Safety Population. Thirteen patients who started had "No study drug administered" and are not included in the Safety Population.
  Among patients in the Safety Population, 67 training phase patients were excluded from efficacy analysis. Completed patients included efficacy phase patients who underwent unenhanced and SonoVue-enhanced ultrasound and had definite truth standard diagnosis available.
Period: Overall Study
Arm/Group | Safety Population
Started | 353
Completed | 259
Not Completed | 94
Not completed — No study drug admimnistered | 13
Not completed — Training Patients | 67
Not completed — No truth standard procedure available | 9
Not completed — Technically inadequate truth standard | 2
Not completed — Indeterminate diagnosis from truth stand | 3

BASELINE CHARACTERISTICS:
Groups:
- ITD Population: All patients who were enrolled in the efficacy phase, received SonoVue, had a definite final diagnosis from truth standard and unenhanced and SonoVue-enhanced ultrasonography available
Arm/Group | ITD Population
Number analyzed (Participants) | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 185
  >=65 years | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 136
Race/Ethnicity, Customized [Number; unit: participants]
  White | 206
  Black | 22
  Asian | 12
  Other | 19
Region of Enrollment [Number; unit: participants]
  United States | 132
  Europe | 93
  Canada | 34

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity: Percentage of True Positive Lesions Among All Malignant Lesions Per Truth Standard
Description: Sensitivity of SonoVue-enhanced ultrasound (SonoVue CE-US) versus unenhanced ultrasound (UE-US) for characterization of malignant focal liver lesions (FLLs) using the diagnosis provided by each of the 3 off-site assessors (blinded to patient data) for the Intent-to-diagnose (ITD) population. Unit of analysis was the lesion, equivalent to subject, since each subject had a single lesion to be characterized.
  True positive: subject with a target lesion characterized as malignant by both ultrasonography and the truth standard.
  Truth standard: CE-CT and/or CE-MRI examination OR tissue pathology/histology from surgical resection/biopsy OR 6-month follow up Calculated as (number of true positive lesions/number of malignant lesions per truth standard) x 100
Time Frame: 24 hours to 6 months
Population: Among 259 ITD subjects, 119 were malignant by truth standard and were included for sensitivity.
Measure: Number (95% Confidence Interval); unit: Percentage of true positive lesions
Units Other Than Participants: Malignant lesions
Groups:
- Offsite Reader 1 UE-US: Offsite Reader 1 UE-US assessment
- Offsite Reader 1 SonoVue CE-US: Offsite Reader 1 SonoVue CE-US assessment
- Offsite Reader 2 UE-US: Offsite Reader 2 UE-US assessment
- Offsite Reader 2 SonoVue CE-US: Offsite Reader 2 SonoVue CE-US assessment
- Offsite Reader 3 UE-US: Offsite Reader 3 UE-US assessment
- Offsite Reader 3 SonoVue CE-US: Offsite Reader 3 SonoVue CE-US assessment
Arm/Group | Offsite Reader 1 UE-US | Offsite Reader 1 SonoVue CE-US | Offsite Reader 2 UE-US | Offsite Reader 2 SonoVue CE-US | Offsite Reader 3 UE-US | Offsite Reader 3 SonoVue CE-US
Number analyzed (Participants) | 119 | 119 | 119 | 119 | 119 | 119
Number analyzed (Malignant lesions) | 119 | 119 | 119 | 119 | 119 | 119
Percentage of true positive lesions | 48.7 [39.8 to 57.7] | 86.6 [80.4 to 92.7] | 35.3 [26.7 to 43.9] | 75.6 [67.9 to 83.3] | 16.0 [9.4 to 22.5] | 91.6 [86.6 to 96.6]
Statistical Analysis 1: Comparison: Offsite Reader 1 UE-US vs Offsite Reader 1 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Sensitivity (%) = 37.8, 95% CI 2-sided [27.4 to 48.2]
Statistical Analysis 2: Comparison: Offsite Reader 2 UE-US vs Offsite Reader 2 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Sensitivity (%) = 40.3, 95% CI 2-sided [30.4 to 50.3]
Statistical Analysis 3: Comparison: Offsite Reader 3 UE-US vs Offsite Reader 3 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Sensitivity (%) = 75.6, 95% CI 2-sided [67.9 to 83.3]

2. Primary Outcome: Specificity: Percentage of True Negative Lesions Among All Benign Lesions Per Truth Standard'
Description: Specificity of SonoVue-enhanced versus unenhanced ultrasound for characterization of benign FLLs, using the diagnosis provided by each of the 3 off-site assessors (blinded to patient data) for the ITD population.
  Unit of analysis was the lesion, equivalent to the subject, since each subject had a single lesion that was to be characterized.
  True negative: subject with a target lesion characterized as benign by both ultrasonography and truth standard.
  Among the 259 ITD participants, only 140 participants (lesions) were benign based on the truth standard.
  Truth standard: CE-CT and /or CE-MRI examination OR tissue pathology/histology from surgical resection/biopsy OR 6-month follow up. Calculated as (number of true negative lesions/number of benign lesions per truth standard) x 100.
Time Frame: 24 hours to 6 months
Population: Among the 259 ITD participants, only 140 participants (lesions) were benign based on the truth standard and were were included for specificty.
Measure: Number (95% Confidence Interval); unit: Percentage of true benign lesions
Units Other Than Participants: Benign lesions
Arm/Group | Offsite Reader 1 UE-US | Offsite Reader 1 SonoVue CE-US | Offsite Reader 2 UE-US | Offsite Reader 2 SonoVue CE-US | Offsite Reader 3 UE-US | Offsite Reader 3 SonoVue CE-US
Number analyzed (Participants) | 140 | 140 | 140 | 140 | 140 | 140
Number analyzed (Benign lesions) | 140 | 140 | 140 | 140 | 140 | 140
Percentage of true benign lesions | 62.9 [54.9 to 70.9] | 70.7 [63.2 to 78.3] | 54.3 [46.0 to 62.5] | 82.9 [76.6 to 89.1] | 22.1 [15.3 to 29.0] | 72.9 [65.5 to 80.2]
Statistical Analysis 1: Comparison: Offsite Reader 1 UE-US vs Offsite Reader 1 SonoVue CE-US; Test type: Superiority or Other; p = 0.1380, McNemar; Difference in Specificity (%) = 7.9, 95% CI 2-sided [-2.4 to 18.2]
Statistical Analysis 2: Comparison: Offsite Reader 2 UE-US vs Offsite Reader 2 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Specificity (%) = 28.6, 95% CI 2-sided [19.7 to 37.5]
Statistical Analysis 3: Comparison: Offsite Reader 3 UE-US vs Offsite Reader 3 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Specificity (%) = 50.7, 95% CI 2-sided [42.0 to 59.5]

3. Secondary Outcome: Accuracy: Percentage of True Positive and True Negative Among All Lesions
Description: Accuracy of SonoVue-enhanced versus unenhanced ultrasound for characterization of malignant and benign FLLs, using the diagnosis provided by each of the 3 off-site assessors (blinded to patient data) for the ITD population.
  Unit of analysis was the lesion, equivalent to the subject, since each subject had a single lesion that was to be characterized.
  True positive: subject with a target lesion characterized as malignant by both ultrasonography and truth standard.
  True negative: subject with a target lesion characterized as benign by both ultrasonography and truth standard.
  Truth standard: CE-CT and /or CE-MRI examination OR tissue pathology/histology from surgical resection/biopsy OR 6-month follow up. Calculated as (number of true positive and true negative lesions/number of total lesions per truth standard) x 100.
Time Frame: 24 hours to 6 months
Population: 259 participants in the ITD population
Measure: Number (95% Confidence Interval); unit: Percent true positive and negative lesio
Units Other Than Participants: Total lesions
Arm/Group | Offsite Reader 1 UE-US | Offsite Reader 1 SonoVue CE-US | Offsite Reader 2 UE-US | Offsite Reader 2 SonoVue CE-US | Offsite Reader 3 UE-US | Offsite Reader 3 SonoVue CE-US
Number analyzed (Participants) | 259 | 259 | 259 | 259 | 259 | 259
Number analyzed (Total lesions) | 259 | 259 | 259 | 259 | 259 | 259
Percent true positive and negative lesio | 56.4 [50.3 to 62.4] | 78.0 [72.9 to 83.0] | 45.6 [39.5 to 51.6] | 79.5 [74.6 to 84.5] | 19.3 [14.5 to 24.1] | 81.5 [76.7 to 86.2]
Statistical Analysis 1: Comparison: Offsite Reader 1 UE-US vs Offsite Reader 1 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Accuracy (%) = 21.6, 95% CI 2-sided [14.1 to 29.2]
Statistical Analysis 2: Comparison: Offsite Reader 2 UE-US vs Offsite Reader 2 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Accuracy (%) = 34.0, 95% CI 2-sided [27.3 to 40.7]
Statistical Analysis 3: Comparison: Offsite Reader 3 UE-US vs Offsite Reader 3 SonoVue CE-US; Test type: Superiority or Other; p < .0001, McNemar; Difference in Accuracy (%) = 75.6, 95% CI 2-sided [67.9 to 83.3]

4. Secondary Outcome: Positive Predictive Value [PPV]: Percentage of True Positive Lesions Among All Malignant Lesions Per Ultrasound
Description: Positive Predictive Value of SonoVue-enhanced versus unenhanced ultrasound for characterization of FLLs, using the diagnosis provided by each of the 3 off-site assessors (blinded to patient data) for the ITD population. Unit of analysis was the lesion, equivalent to the subject, since each subject had a single lesion that was to be characterized.
  True positive: subject with a target lesion characterized as malignant by both ultrasonography and truth standard.
  Truth standard: CE-CT and /or CE-MRI examination OR tissue pathology/histology from surgical resection/biopsy OR 6-month follow up.
  Calculated as (number of true positive lesions/number of malignant lesions per ultrasound) x 100.
Time Frame: 24 hours to 6 months
Population: Among the 259 ITD participants, the overall number of participants (lesions) assessed as malignant varied based on the evaluation of the UE-US and CE-US made by each off-site Reader.
Measure: Number (95% Confidence Interval); unit: Percent positive lesions by ultrasound
Units Other Than Participants: Positive lesions
Arm/Group | Offsite Reader 1 UE-US | Offsite Reader 1 SonoVue CE-US | Offsite Reader 2 UE-US | Offsite Reader 2 SonoVue CE-US | Offsite Reader 3 UE-US | Offsite Reader 3 SonoVue CE-US
Number analyzed (Participants) | 110 | 144 | 106 | 114 | 128 | 147
Number analyzed (Positive lesions) | 110 | 144 | 106 | 114 | 128 | 147
Percent positive lesions by ultrasound | 52.7 [43.4 to 62.1] | 71.5 [64.2 to 78.9] | 39.6 [30.3 to 48.9] | 78.9 [71.5 to 86.4] | 14.8 [8.7 to 21.0] | 74.1 [67.1 to 81.2]
Statistical Analysis 1: Comparison: Offsite Reader 1 UE-US vs Offsite Reader 1 SonoVue CE-US; Test type: Superiority or Other; p < .0001, Wald Test
Statistical Analysis 2: Comparison: Offsite Reader 2 UE-US vs Offsite Reader 2 SonoVue CE-US; Test type: Superiority or Other; p < .0001, Wald Test
Statistical Analysis 3: Comparison: Offsite Reader 3 UE-US vs Offsite Reader 3 SonoVue CE-US; Test type: Superiority or Other; p < .0001, Wald Test

5. Secondary Outcome: Negative Predictive Value [NPV]: Percentage of True Negative Lesions Among All Benign Lesions Per Ultrasound
Description: Negative Predictive Value of SonoVue-enhanced versus unenhanced ultrasound for characterization of FLLs, using the diagnosis provided by each of the 3 off-site assessors (blinded to patient data) for the ITD population. Unit of analysis was the lesion, equivalent to the subject, since each subject had a single lesion that was to be characterized.
  True negative: subject with a target lesion characterized as benign by both ultrasonography and truth standard.
  Truth standard: CE-CT and /or CE-MRI examination OR tissue pathology/histology from surgical resection/biopsy OR 6-month follow up. Calculated as (number of true negative lesions/number of benign lesions per ultrasound) x 100.
Time Frame: 24 hours to 6 months
Population: Among the 259 ITD participants, the number of participants (lesions) assessed as benign varied based on the evaluation of the UE-US and CE-US made by each off-site Reader.
Measure: Number (95% Confidence Interval); unit: Percent negative lesions by ultrasound
Units Other Than Participants: Negative lesions
Arm/Group | Offsite Reader 1 UE-US | Offsite Reader 1 SonoVue CE-US | Offsite Reader 2 UE-US | Offsite Reader 2 SonoVue CE-US | Offsite Reader 3 UE-US | Offsite Reader 3 SonoVue CE-US
Number analyzed (Participants) | 149 | 115 | 153 | 145 | 131 | 112
Number analyzed (Negative lesions) | 149 | 115 | 153 | 145 | 131 | 112
Percent negative lesions by ultrasound | 59.1 [51.2 to 67.0] | 86.1 [79.8 to 92.4] | 49.7 [41.8 to 57.6] | 80.0 [73.5 to 86.5] | 23.7 [16.4 to 30.9] | 91.1 [85.8 to 96.4]
Statistical Analysis 1: Comparison: Offsite Reader 1 UE-US vs Offsite Reader 1 SonoVue CE-US; Test type: Superiority or Other; p < .0001, Wald Test
Statistical Analysis 2: Comparison: Offsite Reader 2 UE-US vs Offsite Reader 2 SonoVue CE-US; Test type: Superiority or Other; p < .0001, Wald Test
Statistical Analysis 3: Comparison: Offsite Reader 3 UE-US vs Offsite Reader 3 SonoVue CE-US; Test type: Superiority or Other; p < .0001, Wald Test

6. Secondary Outcome: Specific Diagnosis of Malignant FLLs
Description: SonoVue-enhanced versus unenhanced ultrasound for specific diagnosis of malignant FLLs, using the diagnosis provided by each of the 3 off-site assessors (blinded to patient data) for the ITD population. Unit of analysis was the lesion, equivalent to the subject, since each subject had a single lesion that was to be characterized.
  Truth standard: CE-CT and /or CE-MRI examination OR tissue pathology/histology from surgical resection/biopsy OR 6-month follow up. Calculated as (number of correctly characterized lesions/number of lesions per truth standard) x 100.
Time Frame: 24 hours to 6 months
Population: Among the 119 ITD participants with malignant lesions based on the truth standard, only 94 participants (lesions) were characterized as either hepatocellular carcinoma (HCC) lesions or metastatic lesions.
Measure: Number; unit: Malignant lesions
Units Other Than Participants: Malignant lesions to be characterized
Arm/Group | Offsite Reader 1 UE-US | Offsite Reader 1 SonoVue CE-US | Offsite Reader 2 UE-US | Offsite Reader 2 SonoVue CE-US | Offsite Reader 3 UE-US | Offsite Reader 3 SonoVue CE-US
Number analyzed (Participants) | 94 | 94 | 94 | 94 | 94 | 94
Number analyzed (Malignant lesions to be characterized) | 94 | 94 | 94 | 94 | 94 | 94
Malignant lesions
  # of HCC by Truth Standard | 47 | 47 | 47 | 47 | 47 | 47
  # HCC(Malignant) Correctly Characterized | 16 | 26 | 10 | 29 | 3 | 30
  # of Metastasis by Truth Standard | 47 | 47 | 47 | 47 | 47 | 47
  # Metastasis Correctly Characterized | 18 | 37 | 12 | 31 | 1 | 28

7. Secondary Outcome: Specific Diagnosis of Benign FLLs
Description: SonoVue-enhanced versus unenhanced ultrasound for specific diagnosis of benign FLLs, using the diagnosis provided by each of the 3 off-site assessors (blinded to patient data) for the ITD population. Unit of analysis was the lesion, equivalent to the subject, since each subject had a single lesion that was to be characterized.
  Among the 140 ITD participants with benign lesions based on the truth standard, only 91 participants (lesions) were characterized as either hemangioma or focal nodular hyperplasia.
  Truth standard: CE-CT and /or CE-MRI examination OR tissue pathology/histology from surgical resection/biopsy OR 6-month follow up. Calculated as (number of correctly characterized lesions/number of lesions per truth standard) x 100.
Time Frame: 24 hours to 6 months
Population: Among the 140 ITD participants with benign lesions based on the truth standard, only 91 participants (lesions) were characterized as either hemangioma or focal nodular hyperplasia.
Measure: Number; unit: Benign lesions
Units Other Than Participants: Benign lesions to be characterized
Arm/Group | Offsite Reader 1 UE-US | Offsite Reader 1 SonoVue CE-US | Offsite Reader 2 UE-US | Offsite Reader 2 SonoVue CE-US | Offsite Reader 3 UE-US | Offsite Reader 3 SonoVue CE-US
Number analyzed (Participants) | 91 | 91 | 91 | 91 | 91 | 91
Number analyzed (Benign lesions to be characterized) | 91 | 91 | 91 | 91 | 91 | 91
Benign lesions
  # of Hemangioma by Truth Standard | 52 | 52 | 52 | 52 | 52 | 52
  # Hemangioma Correctly Characterized | 28 | 38 | 30 | 43 | 12 | 38
  # of Focal nodular hyperplasia by Truth Standard | 39 | 39 | 39 | 39 | 39 | 39
  #Focal nodular hyperplasia Correctly Characterized | 15 | 23 | 8 | 22 | 2 | 18

8. Secondary Outcome: Inter-reader Agreement
Description: Kappa statistic based on assessment of malignant or benign by unenhanced and SonoVue-enhanced ultrasonography separately and computation for the percentage agreement within two categories: "3 out of 3 readers agree" and "2 out of 3 readers agree".
Time Frame: 24 hours to 6 months
Measure: Number; unit: Percentage of agreement
Groups:
- UE-US: UE-US Inter-reader agreement
- CE-US: CE-US Inter-reader agreement
Arm/Group | UE-US | CE-US
Number analyzed (Participants) | 259 | 259
Percentage of agreement
  % Agreement: All 3 off-site readers agree | 28.2 | 66.0
  % Agreement: 2 out of 3 off-site readers agree | 94.6 | 99.6

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of signing the Informed Consent Form through 7 days after SonoVue administration.
Description: An AE was defined as any untoward medical occurrence in a patient or a clinical trial subject administered a medicinal product and that did not necessarily have to have a causal relationship with the use of the product. Any patient who received SonoVue is in the Safety Population.
  Of 353 patients who started the study, 13 had "No study drug administered" and are not included and 340 received SonoVue and are included in the Safety Population.
  All AEs were categorized using MedDRA 12.1.
Groups:
- Safety Population: Interventions included SonoVue administration, unenhanced and SonoVue-enhanced ultrasound and definitive truth standard diagnosis.
  Any patient who received SonoVue, training or efficacy phase, regardless of availability of ultrasonography or truth standard, is included in the Safety Population.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 4/340
Other Adverse Events (participants affected / at risk) | 45/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=340)
Dehydration (Metabolism and nutrition disorders) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=340)
Tinnitus (Ear and labyrinth disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 2
Injection site haemorrhage (General disorders) | 1
Injection site irritation (General disorders) | 1
Injection site pain (General disorders) | 2
Malaise (General disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Basophil count increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results may be presented at scientific symposia or published in a peer-review journal after review by sponsor in accordance with the guidelines set forth in the applicable publication or financial agreement